CLINICAL TRIAL: NCT01984697
Title: A Phase III Clinical Trial to Study the Tolerability and Immunogenicity of a 2-dose Regimen of V503, a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine, Administered in Preadolescents and Adolescents (9 to 14 Year Olds) With a Comparison to Young Women (16 to 26 Year Olds)
Brief Title: A Phase III Study of a 2-dose Regimen of a Multivalent Human Papillomavirus (HPV) Vaccine (V503), Administered to 9 to 14 Year-olds and Compared to Young Women, 16 to 26 Years Old (V503-010)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-010; 2013-001314-15 (EudraCT Number); V503-010 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Girls 9 to 14 Years V503 at Months 0 and 6 (Experimental): Girls aged 9 to 14 years received a 2-dose regimen of V503 0.5 mL intramuscular (IM) injection at Months 0 and 6. An additional dose of V503 0.5 mL IM was administered at Month 36.
  Interventions: Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine)
- Boys 9 to 14 Years V503 at Months 0 and 6 (Experimental): Boys aged 9 to 14 years received a 2-dose regimen of V503 0.5 mL IM injection at Months 0 and 6. An additional dose of V503 0.5 mL IM was administered at Month 36.
  Interventions: Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine)
- Girls and Boys 9 to 14 Years V503 at Months 0 and 12 (Experimental): Girls and boys aged 9 to 14 years received a 2-dose regimen of V503 0.5 mL IM injection at Months 0 and 12. An additional dose of V503 0.5 mL IM was administered at Month 36.
  Interventions: Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine)
- Girls 9 to 14 Years V503 at Months 0, 2, and 6 (Experimental): Girls aged 9 to 14 years received a 3-dose regimen of V503 0.5 mL IM injection at Months 0, 2, and 6. An additional dose of V503 0.5 mL IM was administered at Month 36 for a subset of participants.
  Interventions: Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine)
- Young Women 16 to 26 Years V503 at Months 0, 2, and 6 (Active Comparator): Young Women aged 16 to 26 years received a 3-dose regimen of V503 0.5 mL IM injection at Months 0, 2, and 6. An additional dose of V503 0.5 mL IM was administered at Month 36 for a subset of participants.
  Interventions: Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine)

INTERVENTIONS:
Biological: V503 (9-valent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] vaccine) — V503, a 9-valent HPV (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) administered as a 0.5-mL intramuscular injection

SUMMARY:
This was a 37-month safety and immunogenicity study conducted in boys and girls 9 to 14 years of age and in young women 16 to 26 years of age. From this study, the goal was to establish that the investigational 2-dose regimens (0, 6 months and 0, 12 months) studied in boys and girls 9 to 14 years of age are generally safe and immunogenic, with an antibody response that is not inferior to that observed in young women 16 to 26 years of age who received the standard 3-dose regimen of V503 (i.e., the population and dose regimen used to establish V503 efficacy).

ELIGIBILITY:
Inclusion Criteria:

All Participants:

-Judged to be in good physical health on the basis of medical history, physical examination and laboratory results

Boys and Girls 9 to 14 Years:

-Must not have had coitarche and does not plan on becoming sexually active during the vaccination period

Women 16 to 26 Years:

* Has never had a Papanicolaou (Pap) test or only had normal Pap test results
* A lifetime history of 0 to 4 male and/or female sexual partners

Exclusion Criteria:

All Participants:

* Known allergy to any vaccine component
* History of severe allergic reaction that required medical intervention
* Thrombocytopenia or any coagulation disorder
* Females only: participant is pregnant or expecting to donate eggs during day 1 through month 7
* Currently immunocompromised, or been diagnosed with immunodeficiency
* Had a splenectomy
* Receiving or has received immunosuppressive therapies within the last year
* Received any immunoglobulin product or blood-derived product within 3 months
* Received a marketed HPV vaccine or has participated in an HPV vaccine clinical trial

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1518 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Iversen OE, Miranda MJ, Ulied A, Soerdal T, Lazarus E, Chokephaibulkit K, Block SL, Skrivanek A, Nur Azurah AG, Fong SM, Dvorak V, Kim KH, Cestero RM, Berkovitch M, Ceyhan M, Ellison MC, Ritter MA, Yuan SS, DiNubile MJ, Saah AJ, Luxembourg A. Immunogenicity of the 9-Valent HPV Vaccine Using 2-Dose Regimens in Girls and Boys vs a 3-Dose Regimen in Women. JAMA. 2016 Dec 13;316(22):2411-2421. doi: 10.1001/jama.2016.17615. PMID 27893068
- [Derived] Carter JJ, Smith RA, Scherer EM, Skibinski DAG, Sankaranarayanan S, Luxembourg A, Kollmann T, Marty KD, Sadarangani M, Dobson S, Galloway DA. Term immune memory responses to human papillomavirus (HPV) vaccination following 2 versus 3 doses of HPV vaccine. Vaccine. 2025 Mar 19;50:126817. doi: 10.1016/j.vaccine.2025.126817. Epub 2025 Feb 5. PMID 39914257
- [Derived] Bornstein J, Roux S, Kjeld Petersen L, Huang LM, Dobson SR, Pitisuttithum P, Diez-Domingo J, Schilling A, Ariffin H, Tytus R, Rupp R, Senders S, Engel E, Ferris D, Kim YJ, Tae Kim Y, Kurugol Z, Bautista O, Nolan KM, Sankaranarayanan S, Saah A, Luxembourg A. Three-Year Follow-up of 2-Dose Versus 3-Dose HPV Vaccine. Pediatrics. 2021 Jan;147(1):e20194035. doi: 10.1542/peds.2019-4035. Epub 2020 Dec 22. PMID 33386332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1536 participants were screened and 1518 were randomized into the study.
Period: Overall Study
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Started | 301 | 301 | 301 | 301 | 314
Vaccination 1 | 301 | 301 | 300 | 300 | 314
Vaccination 2 | 293 | 296 | 291 | 298 | 313
Vaccination 3 | 0 | 0 | 0 | 293 | 311
Month 36 Vaccination | 270 | 281 | 280 | 9 | 31
Completed | 258 | 270 | 272 | 280 | 279
Not Completed | 43 | 31 | 29 | 21 | 35
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 14 | 5 | 10 | 6 | 21
Not completed — Physician Decision | 3 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 8 | 5 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 15 | 21 | 13 | 11 | 13
Not completed — Missed last follow-up visit | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6 | Total
Number analyzed (Participants) | 301 | 301 | 301 | 301 | 314 | 1518
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.4 (1.7) | 11.5 (1.7) | 11.4 (1.6) | 11.4 (1.7) | 21.0 (2.7) | 13.4 (4.3)
Age, Customized [Number; unit: Participants]
  Between 9 and 10 years | 100 | 98 | 100 | 101 | 0 | 399
  Between 11 and 12 years | 102 | 102 | 106 | 100 | 0 | 410
  Between 13 and 14 years | 99 | 101 | 95 | 100 | 0 | 395
  Between 16 and 26 years | 0 | 0 | 0 | 0 | 314 | 314
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 0 | 151 | 301 | 314 | 1067
  Male | 0 | 301 | 150 | 0 | 0 | 451

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers to Human Papillomavirus (HPV) Type 6 After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV virus-like particles (VLP) type 6 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: All participants who 1) received all vaccinations in the planned regimen, 2) had a serum sample collected 4 weeks after the last vaccination in the planned regimen, 3) were seronegative at Day 1 for the relevant HPV type, and 4) had no protocol violations that would interfere with evaluation of the immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 258 | 263 | 257 | 254 | 238
mMU/mL | 1657.9 [1479.6 to 1857.6] | 1557.4 [1391.5 to 1743.1] | 2678.8 [2390.2 to 3002.1] | 1496.1 [1334.1 to 1677.8] | 770.9 [684.8 to 867.9]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the Geometric Mean Titer (GMT) ratio for Girls 9 to 14 Years / Young Women 16 to 26 years is >0.67; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.15, 95% CI 2-sided [1.83 to 2.53]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the GMT ratio for Boys 9 to 14 Years / Young Women 16 to 26 years is >0.67; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.02, 95% CI 2-sided [1.73 to 2.36]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the GMT ratio for Girls and Boys 9 to 14 Years / Young Women 16 to 26 years is >0.67; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 3.47, 95% CI 2-sided [2.93 to 4.11]

2. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 6 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 6 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 6 was defined as a titer >=30 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 258 | 263 | 257 | 254 | 238
Percentage of participants | 99.6 [97.9 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 99.2 [97.2 to 99.9] | 99.6 [97.7 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the seroconversion percentage difference for Girls 9 to 14 Years - Young Women 16 to 26 years is > -5; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.0, 95% CI 2-sided [-1.8 to 2.0]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the seroconversion percentage difference for Boys 9 to 14 Years - Young Women 16 to 26 years is > -5; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.3]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the seroconversion percentage difference for Girls and Boys 9 to 14 Years - Young Women 16 to 26 years is > -5; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.1 to 2.3]

3. Primary Outcome: Geometric Mean Titers to HPV Type 11 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 11 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 258 | 264 | 257 | 254 | 238
mMU/mL | 1388.9 [1240.4 to 1555.3] | 1423.9 [1273.2 to 1592.3] | 2941.8 [2626.6 to 3294.9] | 1306.3 [1165.5 to 1464.0] | 580.5 [516.0 to 653.0]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — Non-inferiority is demonstrated if the lower limit of the 95% confidence interval of the GMT ratio for Girls 9 to 14 Years / Young Women 16 to 26 years is >0.67; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.39, 95% CI 2-sided [2.03 to 2.82]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.45, 95% CI 2-sided [2.09 to 2.88]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 5.07, 95% CI 2-sided [4.32 to 5.94]

4. Primary Outcome: Geometric Mean Titers to HPV Type 16 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 16 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 273 | 264 | 269 | 249
mMU/mL | 8004.9 [7160.5 to 8948.8] | 8474.8 [7582.4 to 9472.3] | 14329.3 [12796.4 to 16045.9] | 6996.0 [6254.1 to 7825.8] | 3154.0 [2807.1 to 3543.7]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.54, 95% CI 2-sided [2.14 to 3.00]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.69, 95% CI 2-sided [2.29 to 3.15]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 4.54, 95% CI 2-sided [3.84 to 5.37]

5. Primary Outcome: Geometric Mean Titers to HPV Type 18 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 18 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 272 | 266 | 270 | 267
mMU/mL | 1872.8 [1651.6 to 2123.6] | 1860.9 [1641.1 to 2110.2] | 2810.4 [2474.9 to 3191.3] | 2049.3 [1806.4 to 2324.8] | 761.5 [670.8 to 864.5]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.46, 95% CI 2-sided [2.05 to 2.96]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.44, 95% CI 2-sided [2.04 to 2.92]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 3.69, 95% CI 2-sided [3.06 to 4.45]

6. Primary Outcome: Geometric Mean Titers to HPV Type 31 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 31 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 271 | 268 | 271 | 264
mMU/mL | 1436.3 [1272.1 to 1621.8] | 1498.2 [1326.5 to 1692.0] | 2117.5 [1873.7 to 2393.1] | 1748.3 [1548.1 to 1974.5] | 572.1 [505.8 to 647.2]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.51, 95% CI 2-sided [2.10 to 3.00]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.62, 95% CI 2-sided [2.20 to 3.12]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 3.70, 95% CI 2-sided [3.08 to 4.45]

7. Primary Outcome: Geometric Mean Titers to HPV Type 33 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 33 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 273 | 271 | 269 | 275 | 279
mMU/mL | 1030.0 [920.4 to 1152.7] | 1040.0 [928.9 to 1164.3] | 2197.5 [1961.9 to 2461.3] | 796.4 [712.0 to 890.9] | 348.1 [311.5 to 389.1]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.96, 95% CI 2-sided [2.50 to 3.50]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.99, 95% CI 2-sided [2.55 to 3.50]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 6.31, 95% CI 2-sided [5.36 to 7.43]

8. Primary Outcome: Geometric Mean Titers to HPV Type 45 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 45 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 274 | 273 | 268 | 275 | 280
mMU/mL | 357.6 [313.7 to 407.6] | 352.3 [309.0 to 401.7] | 417.7 [365.9 to 476.9] | 661.7 [580.6 to 754.1] | 213.6 [187.7 to 243.2]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 1.67, 95% CI 2-sided [1.38 to 2.03]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 1.65, 95% CI 2-sided [1.37 to 1.99]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 1.96, 95% CI 2-sided [1.61 to 2.37]

9. Primary Outcome: Geometric Mean Titers to HPV Type 52 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 52 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 273 | 268 | 275 | 271
mMU/mL | 581.1 [521.9 to 647.1] | 640.4 [575.2 to 713.0] | 1123.4 [1008.1 to 1251.9] | 909.9 [817.6 to 1012.5] | 364.2 [327.0 to 405.6]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 1.60, 95% CI 2-sided [1.36 to 1.87]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 1.76, 95% CI 2-sided [1.51 to 2.05]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 3.08, 95% CI 2-sided [2.64 to 3.61]

10. Primary Outcome: Geometric Mean Titers to HPV Type 58 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 58 were measured using a competitive Luminex immunoassay. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 270 | 270 | 265 | 273 | 261
mMU/mL | 1251.2 [1119.6 to 1398.4] | 1325.7 [1186.2 to 1481.6] | 2444.6 [2185.2 to 2734.9] | 1229.3 [1100.7 to 1373.0] | 491.1 [438.6 to 549.8]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT ratio = 2.55, 95% CI 2-sided [2.15 to 3.01]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 2.70, 95% CI 2-sided [2.30 to 3.16]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; p < 0.001, ANOVA; One-sided non-inferiority test at alpha=0.025 level; GMT Ratio = 4.98, 95% CI 2-sided [4.23 to 5.86]

11. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 11 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 11 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 11 was defined as a titer >=16 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 258 | 264 | 257 | 254 | 238
Percentage of participants | 100 [98.6 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 99.6 [97.8 to 100] | 99.6 [97.7 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.1 to 2.3]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.3]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.1 to 2.3]

12. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 16 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 16 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 16 was defined as a titer >=20 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 273 | 264 | 269 | 249
Percentage of participants | 100 [98.7 to 100] | 100 [98.7 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 99.6 [97.8 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.2]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.2]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.2]

13. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 18 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 18 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 18 was defined as a titer >=24 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 272 | 266 | 270 | 267
Percentage of participants | 100 [98.7 to 100] | 100 [98.7 to 100] | 100 [98.6 to 100] | 99.6 [98.0 to 100] | 98.5 [96.2 to 99.6]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 1.5, 95% CI 2-sided [0.1 to 3.8]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 1.5, 95% CI 2-sided [0.1 to 3.8]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 1.5, 95% CI 2-sided [0.1 to 3.8]

14. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 31 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 31 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 31 was defined as a titer >=10 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 271 | 268 | 271 | 264
Percentage of participants | 99.6 [98.0 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 99.6 [97.9 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.0, 95% CI 2-sided [-1.7 to 1.8]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]

15. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 33 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 33 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 33 was defined as a titer >=8 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 273 | 271 | 269 | 275 | 279
Percentage of participants | 99.6 [98.0 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 100 [98.7 to 100] | 99.6 [98.0 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.0, 95% CI 2-sided [-1.7 to 1.7]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.1 to 2.0]

16. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 45 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 45 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 45 was defined as a titer >=8 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 274 | 273 | 268 | 275 | 280
Percentage of participants | 99.3 [97.4 to 99.9] | 99.3 [97.4 to 99.9] | 100 [98.6 to 100] | 99.3 [97.4 to 99.9] | 97.9 [95.4 to 99.2]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 1.4, 95% CI 2-sided [-0.7 to 4.0]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 1.4, 95% CI 2-sided [-0.7 to 4.0]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 2.1, 95% CI 2-sided [0.7 to 4.6]

17. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 52 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 52 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 52 was defined as a titer >=8 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 272 | 273 | 268 | 275 | 271
Percentage of participants | 99.6 [98.0 to 100] | 100 [98.7 to 100] | 100 [98.6 to 100] | 99.6 [98.0 to 100] | 99.6 [98.0 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.0, 95% CI 2-sided [-1.7 to 1.7]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]

18. Secondary Outcome: Percentage of Participants With Seroconversion to HPV Type 58 at Four Weeks After the Last Dose of V503 in the Planned Regimen
Description: Antibodies to HPV VLP type 58 were measured using a competitive Luminex immunoassay. Seroconversion to HPV type 58 was defined as a titer >=8 mMU/mL.
Time Frame: 4 weeks after the last dose of V503 in the planned regimen (Month 7 or Month 13)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 270 | 270 | 265 | 273 | 261
Percentage of participants | 100 [98.6 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 99.6 [98.0 to 100] | 99.6 [97.9 to 100]
Statistical Analysis 1: Comparison: Girls 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]
Statistical Analysis 2: Comparison: Boys 9 to 14 Years V503 at Months 0 and 6 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.0 to 2.1]
Statistical Analysis 3: Comparison: Girls and Boys 9 to 14 Years V503 at Months 0 and 12 vs Young Women 16 to 26 Years V503 at Months 0, 2, and 6; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; p < 0.001, Miettinen and Nurminen; One-sided non-inferiority test at alpha=0.025 level; Seroconversion percentage difference = 0.4, 95% CI 2-sided [-1.1 to 2.1]

19. Other Pre Specified Outcome: Antibody Persistence: Geometric Mean Titers to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 24
Description: Antibodies to HPV VLP types were measured using a competitive Luminex immunoassay. This outcome measure assessed the long-term persistence of antibody response. Antibody titers were expressed as milli Merck units/mL (mMU/mL).
Time Frame: Month 24
Population: All participants who 1) received all vaccinations in the planned regimen, 2) had a serum sample collected 4 weeks after the last vaccination in the planned regimen, 3) were seronegative at Day 1 for the relevant HPV types, and 4) had no protocol violations that would interfere with evaluation of the immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 301 | 301 | 300 | 300 | 314
mMU/mL
  Anti-HPV Type 6: number analyzed (Participants) | 253 | 259 | 252 | 249 | 232
  Anti-HPV Type 6 | 260.7 [231.5 to 293.6] | 209.1 [185.9 to 235.1] | 574.0 [509.6 to 646.5] | 300.7 [266.8 to 339.0] | 153.2 [135.4 to 173.5]
  Anti-HPV Type 11: number analyzed (Participants) | 253 | 260 | 252 | 249 | 232
  Anti-HPV Type 11 | 169.8 [150.5 to 191.7] | 150.6 [133.6 to 169.7] | 443.7 [392.9 to 501.0] | 201.9 [178.7 to 228.1] | 98.3 [86.6 to 111.6]
  Anti-HPV Type 16: number analyzed (Participants) | 266 | 269 | 259 | 264 | 241
  Anti-HPV Type 16 | 900.5 [788.0 to 1028.9] | 801.0 [701.5 to 914.6] | 2316.2 [2023.5 to 2651.4] | 1041.3 [910.8 to 1190.4] | 461.6 [401.2 to 531.0]
  Anti-HPV Type 18: number analyzed (Participants) | 266 | 268 | 261 | 265 | 259
  Anti-HPV Type 18 | 196.8 [174.9 to 221.6] | 169.6 [150.7 to 190.8] | 380.8 [337.9 to 429.1] | 255.8 [227.2 to 288.0] | 122.2 [108.4 to 137.7]
  Anti-HPV Type 31: number analyzed (Participants) | 266 | 267 | 263 | 266 | 258
  Anti-HPV Type 31 | 160.6 [140.8 to 183.3] | 139.1 [122.0 to 158.7] | 312.8 [273.9 to 357.1] | 260.6 [228.4 to 297.3] | 89.6 [78.4 to 102.5]
  Anti-HPV Type 33: number analyzed (Participants) | 267 | 267 | 264 | 270 | 269
  Anti-HPV Type 33 | 131.2 [116.9 to 147.2] | 121.5 [108.3 to 136.4] | 341.7 [304.3 to 383.6] | 120.8 [107.7 to 135.4] | 61.3 [54.6 to 68.7]
  Anti-HPV Type 45: number analyzed (Participants) | 268 | 269 | 263 | 270 | 271
  Anti-HPV Type 45 | 37.8 [33.2 to 43.0] | 31.9 [28.0 to 36.3] | 62.3 [54.7 to 71.1] | 86.9 [76.4 to 98.9] | 30.7 [27.0 to 34.9]
  Anti-HPV Type 52: number analyzed (Participants) | 266 | 269 | 263 | 270 | 261
  Anti-HPV Type 52 | 85.1 [76.4 to 94.7] | 80.9 [72.7 to 90.0] | 199.4 [179.0 to 222.2] | 150.4 [135.2 to 167.4] | 73.7 [66.1 to 82.1]
  Anti-HPV Type 58: number analyzed (Participants) | 264 | 266 | 260 | 268 | 253
  Anti-HPV Type 58 | 155.4 [138.0 to 175.1] | 149.8 [133.1 to 168.6] | 380.2 [337.3 to 428.6] | 183.7 [163.3 to 206.7] | 76.8 [68.0 to 86.7]

20. Other Pre Specified Outcome: Antibody Persistence: Percentage of Participants With Seroconversion to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 24
Description: Antibodies to HPV VLP types were measured using a competitive Luminex immunoassay. This outcome measure assessed the long-term persistence of antibody response. Seroconversion to HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 were defined as a titer >=41, 24, 34, 39, 24, 18, 12, 16, and 12 mMU/mL, respectively. These cutoffs differ from analyses performed on samples collected up to Month 13; the antibody persistence analysis employed a new version of the assay.
Time Frame: Month 24
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 301 | 301 | 300 | 300 | 314
Percentage of participants
  Anti-HPV Type 6: number analyzed (Participants) | 253 | 259 | 252 | 249 | 232
  Anti-HPV Type 6 | 98.4 [96.0 to 99.6] | 96.9 [94.0 to 98.7] | 99.2 [97.2 to 99.9] | 99.6 [97.8 to 100] | 94.0 [90.1 to 96.7]
  Anti-HPV Type 11: number analyzed (Participants) | 253 | 260 | 252 | 249 | 232
  Anti-HPV Type 11 | 98.0 [95.4 to 99.4] | 95.8 [92.6 to 97.9] | 99.6 [97.8 to 100] | 98.8 [96.5 to 99.8] | 94.8 [91.1 to 97.3]
  Anti-HPV Type 16: number analyzed (Participants) | 266 | 269 | 259 | 264 | 241
  Anti-HPV Type 16 | 98.9 [96.7 to 99.8] | 99.6 [97.9 to 100] | 100 [98.6 to 100] | 99.6 [97.9 to 100] | 99.6 [97.7 to 100]
  Anti-HPV Type 18: number analyzed (Participants) | 266 | 268 | 261 | 265 | 259
  Anti-HPV Type 18 | 98.5 [96.2 to 99.6] | 95.9 [92.8 to 97.9] | 98.9 [96.7 to 99.8] | 99.2 [97.3 to 99.9] | 95.0 [91.6 to 97.3]
  Anti-HPV Type 31: number analyzed (Participants) | 266 | 267 | 263 | 266 | 258
  Anti-HPV Type 31 | 97.0 [94.2 to 98.7] | 94.8 [91.4 to 97.1] | 98.5 [96.2 to 99.6] | 97.7 [95.2 to 99.2] | 91.5 [87.4 to 94.6]
  Anti-HPV Type 33: number analyzed (Participants) | 267 | 267 | 264 | 270 | 269
  Anti-HPV Type 33 | 97.8 [95.2 to 99.2] | 96.6 [93.7 to 98.4] | 99.2 [97.3 to 99.9] | 98.9 [96.8 to 99.8] | 94.8 [91.4 to 97.1]
  Anti-HPV Type 45: number analyzed (Participants) | 268 | 269 | 263 | 270 | 271
  Anti-HPV Type 45 | 88.4 [84.0 to 92.0] | 85.9 [81.1 to 89.8] | 93.9 [90.3 to 96.5] | 96.7 [93.8 to 98.5] | 82.7 [77.6 to 87.0]
  Anti-HPV Type 52: number analyzed (Participants) | 266 | 269 | 263 | 270 | 261
  Anti-HPV Type 52 | 96.6 [93.7 to 98.4] | 95.2 [91.9 to 97.4] | 99.2 [97.3 to 99.9] | 99.3 [97.3 to 99.9] | 97.3 [94.6 to 98.9]
  Anti-HPV Type 58: number analyzed (Participants) | 264 | 266 | 260 | 268 | 253
  Anti-HPV Type 58 | 98.9 [96.7 to 99.8] | 99.6 [97.9 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100] | 96.0 [92.9 to 98.1]

21. Other Pre Specified Outcome: Antibody Persistence: Geometric Mean Titers to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 36
Description: as for outcome 19
Time Frame: Month 36
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 301 | 301 | 300 | 300 | 314
mMU/mL
  Anti-HPV Type 6: number analyzed (Participants) | 236 | 254 | 246 | 240 | 214
  Anti-HPV Type 6 | 209.6 [184.9 to 237.6] | 160.1 [141.9 to 180.7] | 401.2 [354.8 to 453.7] | 232.2 [205.1 to 263.0] | 133.8 [117.3 to 152.7]
  Anti-HPV Type 11: number analyzed (Participants) | 236 | 255 | 246 | 240 | 214
  Anti-HPV Type 11 | 133.7 [117.6 to 152.1] | 115.2 [101.8 to 130.3] | 308.2 [271.8 to 349.6] | 159.1 [140.0 to 180.7] | 82.9 [72.4 to 94.9]
  Anti-HPV Type 16: number analyzed (Participants) | 248 | 263 | 253 | 255 | 222
  Anti-HPV Type 16 | 673.8 [582.8 to 779.1] | 592.6 [514.7 to 682.4] | 1534.3 [1328.8 to 1771.5] | 792.4 [686.7 to 914.4] | 368.9 [316.4 to 430.0]
  Anti-HPV Type 18: number analyzed (Participants) | 248 | 262 | 255 | 256 | 239
  Anti-HPV Type 18 | 158.9 [140.8 to 179.4] | 141.7 [125.9 to 159.4] | 276.4 [245.3 to 311.6] | 206.5 [183.3 to 232.7] | 104.1 [92.0 to 117.8]
  Anti-HPV Type 31: number analyzed (Participants) | 248 | 261 | 257 | 258 | 235
  Anti-HPV Type 31 | 127.8 [111.4 to 146.5] | 106.9 [93.5 to 122.1] | 218.0 [190.6 to 249.4] | 205.9 [180.0 to 235.5] | 74.6 [64.8 to 85.9]
  Anti-HPV Type 33: number analyzed (Participants) | 249 | 261 | 258 | 261 | 246
  Anti-HPV Type 33 | 106.0 [94.1 to 119.5] | 95.7 [85.1 to 107.5] | 240.4 [213.8 to 270.3] | 95.5 [85.0 to 107.3] | 52.2 [46.3 to 58.9]
  Anti-HPV Type 45: number analyzed (Participants) | 250 | 263 | 257 | 261 | 248
  Anti-HPV Type 45 | 30.6 [26.9 to 35.0] | 26.8 [23.6 to 30.4] | 43.6 [38.3 to 49.7] | 66.1 [58.1 to 75.2] | 27.3 [23.9 to 31.1]
  Anti-HPV Type 52: number analyzed (Participants) | 248 | 263 | 257 | 261 | 239
  Anti-HPV Type 52 | 66.2 [59.1 to 74.0] | 63.4 [56.8 to 70.7] | 143.2 [128.3 to 159.9] | 115.9 [103.9 to 129.3] | 61.5 [54.8 to 68.9]
  Anti-HPV Type 58: number analyzed (Participants) | 246 | 261 | 255 | 259 | 231
  Anti-HPV Type 58 | 125.8 [111.1 to 142.5] | 119.2 [105.6 to 134.5] | 265.3 [234.8 to 299.8] | 143.0 [126.7 to 161.5] | 64.7 [56.9 to 73.6]

22. Other Pre Specified Outcome: Antibody Persistence: Percentage of Participants With Seroconversion to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 36
Description: as for outcome 20
Time Frame: Month 36
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
Number analyzed (Participants) | 301 | 301 | 300 | 300 | 314
Percentage of participants
  Anti-HPV Type 6: number analyzed (Participants) | 236 | 254 | 246 | 240 | 214
  Anti-HPV Type 6 | 95.3 [91.8 to 97.7] | 91.3 [87.2 to 94.5] | 99.2 [97.1 to 99.9] | 97.9 [95.2 to 99.3] | 92.1 [87.6 to 95.3]
  Anti-HPV Type 11: number analyzed (Participants) | 236 | 255 | 246 | 240 | 214
  Anti-HPV Type 11 | 94.1 [90.2 to 96.7] | 92.9 [89.1 to 95.8] | 99.2 [97.1 to 99.9] | 98.8 [96.4 to 99.7] | 92.1 [87.6 to 95.3]
  Anti-HPV Type 16: number analyzed (Participants) | 248 | 263 | 253 | 255 | 222
  Anti-HPV Type 16 | 97.2 [94.3 to 98.9] | 98.5 [96.2 to 99.6] | 100 [98.6 to 100] | 99.2 [97.2 to 99.9] | 98.2 [95.5 to 99.5]
  Anti-HPV Type 18: number analyzed (Participants) | 248 | 262 | 255 | 256 | 239
  Anti-HPV Type 18 | 95.6 [92.2 to 97.8] | 94.3 [90.7 to 96.8] | 97.6 [94.9 to 99.1] | 97.3 [94.4 to 98.9] | 90.8 [86.4 to 94.1]
  Anti-HPV Type 31: number analyzed (Participants) | 248 | 261 | 257 | 258 | 235
  Anti-HPV Type 31 | 94.0 [90.2 to 96.6] | 91.2 [87.1 to 94.3] | 96.5 [93.5 to 98.4] | 97.7 [95.0 to 99.1] | 86.0 [80.8 to 90.1]
  Anti-HPV Type 33: number analyzed (Participants) | 249 | 261 | 258 | 261 | 246
  Anti-HPV Type 33 | 94.0 [90.3 to 96.6] | 96.9 [94.1 to 98.7] | 99.2 [97.2 to 99.9] | 98.1 [95.6 to 99.4] | 91.9 [87.7 to 95.0]
  Anti-HPV Type 45: number analyzed (Participants) | 250 | 263 | 257 | 261 | 248
  Anti-HPV Type 45 | 83.6 [78.4 to 88.0] | 81.4 [76.1 to 85.9] | 87.9 [83.3 to 91.7] | 91.2 [87.1 to 94.3] | 77.8 [72.1 to 82.8]
  Anti-HPV Type 52: number analyzed (Participants) | 248 | 263 | 257 | 261 | 239
  Anti-HPV Type 52 | 93.5 [89.7 to 96.3] | 93.9 [90.3 to 96.5] | 98.8 [96.6 to 99.8] | 97.7 [95.1 to 99.2] | 95.0 [91.4 to 97.4]
  Anti-HPV Type 58: number analyzed (Participants) | 246 | 261 | 255 | 259 | 231
  Anti-HPV Type 58 | 98.0 [95.3 to 99.3] | 99.2 [97.3 to 99.9] | 100 [98.6 to 100] | 98.8 [96.7 to 99.8] | 94.8 [91.1 to 97.3]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: Up to Month 37; Non-injection site adverse events: up to Day 15 following any vaccination; Injection site adverse events: up to Day 5 following any vaccination
Description: Participants at risk for adverse events includes those who were vaccinated and had safety follow-up data
Arm/Group | Girls 9 to 14 Years V503 at Months 0 and 6 | Boys 9 to 14 Years V503 at Months 0 and 6 | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 | Girls 9 to 14 Years V503 at Months 0, 2, and 6 | Young Women 16 to 26 Years V503 at Months 0, 2, and 6
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/296 | 0/293 | 1/300 | 0/313
Serious Adverse Events (participants affected / at risk) | 6/294 | 9/296 | 6/293 | 6/300 | 11/313
Other Adverse Events (participants affected / at risk) | 53/294 | 32/296 | 46/293 | 55/300 | 90/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Girls 9 to 14 Years V503 at Months 0 and 6 (N=294) | Boys 9 to 14 Years V503 at Months 0 and 6 (N=296) | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 (N=293) | Girls 9 to 14 Years V503 at Months 0, 2, and 6 (N=300) | Young Women 16 to 26 Years V503 at Months 0, 2, and 6 (N=313)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Girls 9 to 14 Years V503 at Months 0 and 6 (N=294) | Boys 9 to 14 Years V503 at Months 0 and 6 (N=296) | Girls and Boys 9 to 14 Years V503 at Months 0 and 12 (N=293) | Girls 9 to 14 Years V503 at Months 0, 2, and 6 (N=300) | Young Women 16 to 26 Years V503 at Months 0, 2, and 6 (N=313)
Injection site pain (General disorders) | 49 (65) | 28 (31) | 41 (52) | 53 (81) | 80 (148)
Headache (Nervous system disorders) | 8 (9) | 9 (9) | 7 (8) | 7 (8) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.